CLINICAL TRIAL: NCT00443170
Title: A Randomized, Blinded, Placebo-controlled Study to Investigate the Safety, and Pharmacokinetics of Single and Repeat Dose Escalation of the Oral YAK3/DYRK3 Inhibitor GSK626616AC in Healthy Subjects
Brief Title: A Placebo-controlled Study to Investigate the Safety, and Pharmacokinetics of Oral GSK626616AC in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: YAK106752
Record Dates: First submitted 2007-03-01; First posted 2007-03-05 (Estimated); Last update posted 2012-03-19 (Estimated); Status verified 2011-02

CONDITIONS: Healthy Subjects; Anaemia
Keywords: repeat dose,; GSK626616AC,; pharmacokinetic,; single dose,; cytochrome P450,; First time in human,; healthy volunteers
MeSH Terms: conditions — Anemia | interventions — Midazolam; Omeprazole; Caffeine; Flurbiprofen; Rosiglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: GSK626616, placebo, midazolam
Drug: omeprazole, caffeine, flurbiprofen, rosiglitazone
  Other Names: omeprazole; caffeine; flurbiprofen; rosiglitazone; GSK626616; placebo; midazolam

SUMMARY:
This is a first time in human study to investigate the safety of GSK626616AC given as oral single and repeat doses in healthy subjects. An additional group of subjects will be assessed to determine the effect of several drugs given at the same time as GSK626616.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 55 years healthy subjects
* Hemoglobin values of 13.5-17.0 g/dL for males or 12.0-15.5 g/dL for females.
* Females cannot be pregnant.

Exclusion Criteria:

* Cannot have exposure to greater than 4 new chemical entities within 12 months.
* Cannot have a clinical history of current alcohol, or illicit drug use which, in the judgment of the Investigator, would interfere with the subject's ability to comply with the dosing schedule.
* Cannot have a history of regular use of tobacco- or nicotine-containing products within 3 months.
* Must not have received a blood transfusion or had a donation of blood within 3 months prior to study entry.
* Cannot use be taking prescription, non-prescription or illicit drugs.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2006-11

PRIMARY OUTCOMES:
adverse events at end of each cohort | end of each cohort
hematology/chemistry/urinalysis at end of each cohort | end of each cohort
physical examination at end of each cohort | end of each cohort
vital signs and electrocardiogram (ECG) at end of each cohort | end of each cohort

SECONDARY OUTCOMES:
GSK626616 pharmacokinetics at end of each cohort | end of each cohort
hemoglobin at end of each cohort | end of each cohort
red blood cell measurements at end of each cohort | end of each cohort
estimates of CYP enzyme activity at end of study | end of study
mRNA levels in peripheral blood at end of study | end of study

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- Australia (3):
  - GSK Investigational Site, Randwick, Sydney, New South Wales
  - GSK Investigational Site, Herston, Queensland
  - GSK Investigational Site, Adelaide, South Australia